CLINICAL TRIAL: NCT04871945
Title: Evaluation of Protective Antibody Production After COVID-19 Vaccination Among Patients Under Hemodialysis
Brief Title: Protective Antibody Level After COVID-19 Vaccination Among Patients Under Hemodialysis
Status: Completed | Type: Observational
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Seegene Medical Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-02-033
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Vaccine Reaction; Hemolysis; End-stage Renal Disease
MeSH Terms: conditions — COVID-19; Hemolysis; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Elecsys Anti-SARS-CoV-2 S (Roche Diagnostics GmbH, Mannheim, Germany), 2) ACCESS SARS-CoV-2 IgG II (Beckman Coulter, Inc. USA) — The antibody level will be measured by the above mentioned methods. The trial drugs are not used but the vaccine that included in National Immunization Program for COVID-19 in Korea will be used for the study.

SUMMARY:
The aim of the study is to evaluate the level of neutralizing antibody against SARS-CoV-2 after COVID-19 vaccination in patients under hemodialysis. To this end, the level of neutralizing antibody of patients under hemodialysis is compared to that of healthy population.

ELIGIBILITY:
Inclusion Criteria:

* The person who is vaccinated with ChAdOx1 (COVID-19 vaccine)
* The person who agrees with the protocol of the study

Exclusion Criteria:

* Age < 18 years
* Pregnants
* Experience of COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients group : Patients under hemodialysis Control group : Healthy population
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
The change in the level of neutralizing antibody against SARS-CoV-2 | Day 0, 14, 28, 56, 91, 120

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park JS, Minn D, Hong S, Jeong S, Kim S, Lee CH, Kim B. Immunogenicity of COVID-19 Vaccination in Patients With End-Stage Renal Disease Undergoing Maintenance Hemodialysis: The Efficacy of a Mix-and-Match Strategy. J Korean Med Sci. 2022 Jun 13;37(23):e180. doi: 10.3346/jkms.2022.37.e180. PMID 35698835